CLINICAL TRIAL: NCT01838772
Title: Effectiveness and Tolerability of Hepatitis C Treatment in HIV Co-infected Patients in Routine Care Services in Asia: A Pilot Model of Care Project
Brief Title: HCV Treatment in HIV Co-Infected Patients in Asia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: amfAR, The Foundation for AIDS Research (Other)
Collaborators: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA010
Record Dates: First submitted 2013-04-05; First posted 2013-04-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C; HIV
Keywords: HCV and HIV co-infection
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegylated-Interferon and Ribavirin (Other): Pegylated-interferon 1.5 microgr/kg, subcutaneously, once weekly for 48 weeks*. Ribavirin, weight-based dosage, divided in two daily doses for 48 weeks*.
  *patients with genotype 2 and 3, moderate liver fibrosis, and rapid virologic response will receive therapy for 24 weeks.
  Interventions: Drug: Pegylated-Interferon and Ribavirin

INTERVENTIONS:
Drug: Pegylated-Interferon and Ribavirin — This is an open-label, single arm demonstration study. Intervention consists in treatment with Pegylated-interferon (Peg-Intron®, 1.5 microgr/kg/week, as subcutaneous injection) and ribavirin (Rebetol®, weight-based dosing, 2-daily doses) for 48 weeks, or 24 weeks for patients with genotype 2 and 3, moderate liver fibrosis, and rapid virological response.
  Other Names: PegIntron; Rebetol

SUMMARY:
The purpose of this study is to assess the effectiveness and tolerability of hepatitis C virus (HCV) treatment in HIV co-infected patients in routine health care services in Asia through a pilot model of care for treatment of HCV in resource-limited settings.

DETAILED DESCRIPTION:
It is estimated that 130-170 million people are chronically infected with the hepatitis C virus (HCV). Out of the 33 million HIV-infected people around the world, it is estimated that at least 5 million are also infected with HCV. HCV therapy with Pegylated-interferon and ribavirin is between 50-90% effective to achieve cure, depending on the virus genotype and patient characteristics, such as ethnicity and IL28B polymorphism. Treatment studies in HIV-uninfected populations have shown that Asian patients experience higher treatment response rates than Caucasians. Unfortunately, although HCV therapy is routinely offered in resource-rich settings, it is essentially inaccessible in resource-limited settings (RLS), where most of the people infected with the virus live. One of the bottlenecks to increasing implementation of HCV therapy in RLS is that therapy is currently expensive and deemed complex for broad implementation in RLS. Through this project and study, TREAT Asia aims to build a regional approach in Asia to establish the feasibility of HCV therapy in HIV-infected patients in RLS, and implement an innovative model of HCV-HIV care that can be expanded in the future.

Patients with HIV infection and documented HCV antibodies under routine HIV care at the four study sites will have HCV RNA testing. Patients with confirmed chronic HCV infection will have HCV genotype and IL28B testing, as well as liver disease assessment with Fibroscan®. Patients with chronic HCV co-infection with any genotype and meeting all other treatment eligibility criteria will be offered treatment with pegylated-interferon and ribavirin through an open-label single arm study. A total of up to 200 patients will be enrolled into the study. Patients will receive intensive treatment preparedness counseling, and ongoing treatment adherence support. Most patients will receive treatment for a total of 48 weeks, but patients with HCV genotype 2 and 3, moderate liver fibrosis, and rapid virological response (negative HCV RNA by four weeks of therapy) will receive 24 weeks of therapy. The primary endpoint of interest will be the proportion of patients achieving sustained virological response, defined as an undetectable HCV RNA 24 weeks after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed HIV infection by antibody and/or virologic testing
* Chronic HCV infection with any genotype, confirmed by a positive anti-HCV antibody test obtained at least six months prior to screening, and detectable HCV RNA at screening.
* Stable ART in patients with CD4 counts between 200-350 cells/µl at the time of screening, OR stable ART, or no ART in patients with CD4 counts above 350 cells/µl at the time of screening.
* Liver fibrosis stage >F1 (defined as a fibrosis score >=7.5 KPa by Fibroscan®, or through histological examination of a liver biopsy specimen).
* Compensated liver disease, with a Child-Pugh grade no greater than A, and:
* No ascites (current or ever)
* No hepatic encephalopathy (current or ever)
* No bleeding varices (current or ever)
* Patients with suspected cirrhosis (Fibroscan® >=13.0 KPa or through histological examination of a liver biopsy specimen) must have an abdominal ultrasound and alpha fetoprotein test result without evidence of hepatocellular carcinoma within two months prior to screening.
* Negative urine or blood pregnancy test for women of childbearing potential documented within the 24-hour period prior to the first dose of study drug.
* All males and females of reproductive age and potential must agree to use effective contraception during treatment and during the 24 weeks after the end of treatment.
* Voluntarily signed informed consent form.
* Willingness to start therapy and to adhere to the requirements of the study visits schedule.

Exclusion Criteria:

* Any history of previous Interferon or ribavirin therapy.
* Known active bacterial infection.
* Ongoing treatment for mycobacterial infection.
* CD4 count <200 cells/ µl.
* Current pregnancy or breast feeding.
* Male partners of women who are pregnant.
* Evidence of a medical condition other than HCV identified as another significant cause of chronic liver disease (e.g., severe alcoholic liver disease, toxin exposures, metabolic liver disease, autoimmune hepatitis).
* Active drug use or alcohol consumption that is judged by the study physician to potentially compromise treatment safety.
* Hemoglobin <11 g/dL in women or <12 g/dL in men.
* ALT (SGPT) or AST (SGOT) level >10 times the upper normal limit.
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3.
* Serum creatinine level >1.5 times the upper normal limit.
* Inadequately controlled thyroid dysfunction (i.e., TSH and T4 levels out of normal ranges).
* Ongoing severe psychiatric disease (e.g., depression) as judged by the study physician to potentially compromise treatment safety.
* Uncontrolled seizure disorder.
* Concomitant use of didanosine.
* Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension.
* History of severe chronic pulmonary disease, cardiac disease, malignancy, or other severe illness, which would make the patient, in the opinion of the study physician, unsuitable for treatment administration and participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with sustained virological response (SVR), defined as an undetectable HCV RNA, 24 weeks after completion of therapy | 24 weeks after completion of therapy

SECONDARY OUTCOMES:
Proportion of patients with Rapid Virological Response (RVR) | 4 weeks of therapy
Proportion of patients with Early Virological Response (EVR) | 12 weeks of therapy
Proportion of patients with End of Treatment Response (ETR) | Up to 48 weeks of therapy
Proportions of patients who discontinue treatment prematurely | Up to 48 weeks of therapy
Clinical and laboratory safety parameters | Up to 48 weeks of therapy
  The proportion of participants with all grades of adverse events will be summarized by severity and relation to study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Durier, MD, MPH, Principal Investigator — TREAT Asia/ amfAR - The Foundation for AIDS Research; Gail Matthews, MD, PhD, Principal Investigator — Kirby Institute
Locations (4):
- Cipto Mangunkusumo General Hospital, Jakarta, Indonesia
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- HIV-NAT/ Thai Red Cross AIDS Research Center, Bangkok, Thailand
- National Hospital for Tropical Diseases, Hanoi, Vietnam